CLINICAL TRIAL: NCT00623233
Title: A Phase 2 Study of Gemcitabine and Bevacizumab as First-Line Treatment in HER2 Negative, Locally Recurrent or Metastatic Breast Cancer Previously Treated With Taxanes
Brief Title: Gemcitabine Plus Bevacizumab in Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11649; B9E-US-S379 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2011-12

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer
Keywords: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Bevacizumab (Experimental): Gemcitabine 2500 milligrams per square meter (mg/m^2) intravenous (IV) over 30 minutes given on Day 1 every 14 days (q 14 days) until disease progression (PD) or unacceptable toxicity.
  Bevacizumab 10 milligrams per kilogram (mg/kg) initially over 90 minutes given on Day 1 q 14 days until PD or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 2500 mg/m^2 IV over 30 minutes given on Day 1 q 14 days prior to bevacizumab until PD or unacceptable toxicity.
  Other Names: Gemzar; LLY188011
Drug: Bevacizumab — Bevacizumab 10 mg/kg IV over 90 minutes at Cycle 1; infusion time may have been decreased for subsequent cycles. (For example, if the first infusion was tolerated without an infusion-associated adverse event [AE], the second infusion was delivered over 60 minutes. If the 60-minute infusion was well tolerated, all subsequent infusions were delivered over 30 minutes.)
  Bevacizumab 10 mg/kg initially over 90 minutes given on Day 1 q 14 days until PD or unacceptable toxicity.

SUMMARY:
To determine how long Gemcitabine and Bevacizumab will stop the cancer from growing in patients with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must be female and greater than or equal to 18 yrs of age
* Participants must have confirmed cancer with measurable or evaluable, locally recurrent or metastatic disease.
* Participants must have received a taxane as neo-adjuvant and/or adjuvant therapy
* Participants may have received prior hormone therapy for locally recurrent or metastatic disease

Exclusion Criteria:

* Participants with breast cancer overexpressing Human Epidermal growth factor Receptor 2 (HER2) gene amplification
* Prior chemotherapy or targeted therapy for metastatic breast cancer
* Prior treatment with gemcitabine, trastuzumab, lapatinib or bevacizumab in any setting
* History of, or active brain mets
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to treatment, or anticipation of need for major surgical procedure during course of study
* Prior history of high blood pressure crisis
* Have a serious, nonhealing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longmont, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfield, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lambertville, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Falls, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Germantown, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport News, Virginia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg: Gemcitabine 2500 milligrams per square meter (mg/m^2) intravenous (IV) over 30 minutes given on Day 1 every 14 days (q 14 days) until disease progression (PD) or unacceptable toxicity.
  Bevacizumab 10 milligrams per kilogram (mg/kg) initially over 90 minutes given on Day 1 q 14 days until PD or unacceptable toxicity.
Period: Overall Study
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Started | 52
Completed | 28 (Included those who discontinued due to PD or death and those who achieved complete response (CR).)
Not Completed | 24
Not completed — Adverse Event | 10
Not completed — Physician Decision | 10
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African descent | 11
  Caucasian | 41
Region of Enrollment [Number; unit: participants]
  United States | 52
Estrogen Receptor (ER) Status [Number; unit: participants] — ER status was used at baseline as a descriptor of the breast cancer tumor population that was studied. ER status had prognostic and treatment implications that made reporting of this characteristic medically relevant.
  participants
    ER+ | 33
    ER- | 19
Progesterone Receptor (PR) Status [Number; unit: participants] — PR status was used at baseline as a descriptor of the breast cancer tumor population that was studied. PR status had prognostic and treatment implications that made reporting of this characteristic medically relevant.
  participants
    PR+ | 30
    PR- | 22
Human Epidermal Growth Factor Receptor 2 (HER2/neu) [Number; unit: participants] — HER2/neu status was used at baseline as a descriptor of the breast cancer tumor population that was studied. HER2/neu status had prognostic and treatment implications that made reporting of this characteristic medically relevant. Breast cancer participants with HER2/neu immunohistochemistry (IHC) 2+ were tested using fluorescence in situ hybridization (FISH). Participants who overexpressed HER2 gene amplication by way of FISH or overexpressed IHC 3+ were not eligible.
  participants
    HER2/neu+ | 0
    HER2/neu- | 52
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classified participants according to their functional impairment. Scores ranged from 0-5: 0=Fully Active; 1=Ambulatory, Restricted Strenuous Activity; 2=Ambulatory, No Work Activities; 3=Partially Confined to Bed, Limited Self Care; 4=Completely Disabled; 5=Death.
  participants
    0 | 28
    1 | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Time
Description: PFS was measured from date of first dose to first date of progressive disease (PD) or death from any cause. For each participant who was not known to have died or to have had PD as of the data inclusion cut-off date for a particular analysis, PFS duration was censored for that analysis at the date of the participant's last progression-free tumor assessment before that cut-off date.
Time Frame: Baseline to measured PD or death from any cause. Tumor assessments were performed every 8 weeks during therapy and every 2 months during post-therapy until documented PD (up to 34 months).
Population: The intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study drug. Participants with events=41; censored participants=11.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 52
months | 4.80 [3.42 to 7.56]

2. Secondary Outcome: Overall Tumor Response Rate (ORR)
Description: Response defined per Response Evaluation Criteria In Solid Tumors (RECIST) criteria: complete response (CR)=disappearance of all target lesions; partial response (PR)=30% decrease in sum of longest diameter of target lesions; progressive disease (PD)=20% increase in sum of longest diameter of target lesions; stable disease=small changes that do not meet above criteria. ORR=proportion of participants who achieved a confirmed best response of CR or PR (responders). ORR=number of participants with CR or PR /number of participants qualified for tumor response analysis (per protocol population).
Time Frame: Baseline to measured PD. Tumor assessments were performed every 8 weeks (q 8 weeks) during therapy and q 2 months during post-therapy until documented PD (up to 34 months).
Population: The per protocol (PP) population included all intent-to-treat (ITT) participants who met the following criteria: histological or cytological diagnosis of breast cancer; presence of measurable disease at baseline per RECIST criteria; had at least 1 dose of study drug; no current systemic anti-tumor treatment other than protocol-specified therapy.
Measure: Number (95% Confidence Interval); unit: proportion of responders
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 42
proportion of responders | 0.214 [0.1030 to 0.3681]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs); Pharmacology Toxicities
Description: A listing of serious adverse events (SAEs) and other non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Baseline, every cycle (every 14 days) up to 34 months
Population: The safety population was the treated population and included all participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 52
participants
  SAEs | 18
  Other non-serious AEs | 51

4. Secondary Outcome: 1-Year Overall Survival (OS) Rate
Description: OS was measured from the date of first dose to the date of death from any cause. For each participant who was not known to have died as of the data inclusion cut-off date for a particular analysis, OS duration was censored for that analysis at the date of participant's last study contact prior to that cut-off date. The 1-year survival rate (percentage of participants who were alive at 1 year) was estimated from OS data.
Time Frame: Baseline to death from any cause, 1 year
Population: The intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study drug. Participants with events=25; censored participants=27.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 52
percentage of participants | 68.68 [54.05 to 79.50]

ADVERSE EVENTS:
Arm/Group | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 18/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg (N=52)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4)
Asthenia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin Infection (Infections and infestations) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fluid Retention (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2)
Head Discomfort (Nervous system disorders) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 1 (1)
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine 2500 mg/m^2 + Bevacizumab 10 mg/kg (N=52)
Anaemia (Blood and lymphatic system disorders) | 16 (18)
Leukopenia (Blood and lymphatic system disorders) | 10 (14)
Neutropenia (Blood and lymphatic system disorders) | 14 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (12)
Sinus Tachycardia (Cardiac disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 6 (7)
Abdominal Pain (Gastrointestinal disorders) | 6 (6)
Abdominal Pain Lower (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 21 (22)
Diarrhoea (Gastrointestinal disorders) | 12 (18)
Dyspepsia (Gastrointestinal disorders) | 7 (10)
Nausea (Gastrointestinal disorders) | 32 (51)
Stomatitis (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 14 (17)
Asthenia (General disorders) | 4 (4)
Chest Pain (General disorders) | 3 (4)
Fatigue (General disorders) | 32 (38)
Influenza Like Illness (General disorders) | 3 (4)
Oedema (General disorders) | 4 (5)
Oedema Peripheral (General disorders) | 4 (4)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 7 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 7 (7)
Alanine Aminotransferase Increased (Investigations) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 3 (4)
Blood Alkaline Phosphatase Increased (Investigations) | 3 (3)
Weight Decreased (Investigations) | 5 (5)
Decreased Appetite (Metabolism and nutrition disorders) | 15 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 11 (13)
Neuropathy Peripheral (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 6 (7)
Insomnia (Psychiatric disorders) | 4 (5)
Proteinuria (Renal and urinary disorders) | 13 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Hypertension (Vascular disorders) | 12 (16)
Lymphoedema (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days